CLINICAL TRIAL: NCT02953821
Title: A Multicenter, Randomized, Double Blind, Placebo Controlled Study to Assess the Efficacy and Safety of Acthar Gel in Subjects With Persistently Active Systemic Lupus Erythematosus Despite Moderate Dose Corticosteroids
Brief Title: Acthar Gel for Active Systemic Lupus Erythematosus (SLE)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MNK14304067
Record Dates: First submitted 2016-11-01; First posted 2016-11-03 (Estimated); Results first posted 2020-08-20 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Lupus Erythematosus, Systemic
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acthar Gel (Experimental): Participants receive Acthar Gel every other day for 4 weeks, and then twice per week for 20 weeks
  Interventions: Drug: Acthar Gel
- Placebo Gel (Placebo Comparator): Participants receive Placebo Gel every other day for 4 weeks, and then twice per week for 20 weeks
  Interventions: Drug: Placebo Gel

INTERVENTIONS:
Drug: Acthar Gel — 1 mL (80 Units) given by a shot under the skin (via subcutaneous injection)
  Other Names: Repository corticotropin
  Arms: Acthar Gel
Drug: Placebo Gel — 1 mL (0 Units) given by a shot under the skin (via subcutaneous injection)
  Other Names: Matching placebo
  Arms: Placebo Gel

SUMMARY:
This trial is to study Acthar Gel in participants with active systemic lupus erythematosus (SLE).

The doctor will assign eligible patients to one of two groups (like flipping a coin).

Participants will receive the treatment assigned to their group for 24 weeks:

* Acthar Gel
* Placebo Gel, which looks like Acthar Gel, but has no medicine in it.

The doctor or his staff will take measurements and ask questions to:

* see how well the gel is working
* see how safe it is for patients with SLE

DETAILED DESCRIPTION:
This trial was initiated (started recruiting) in October 2016, but first patient was not enrolled (randomized) until December, 2016.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate in this trial, a patient must:

* Have a diagnosis of SLE according to 4 of the American College of Rheumatology revised criteria
* Have active SLE
* Have moderate to severe rash and/or arthritis as demonstrated by BILAG-2004 score A or B in the mucocutaneous and/or musculoskeletal body systems at both Screening and Randomization Visits
* Have a documented history or screening result of

  1. positive antinuclear antibody (ANA), OR
  2. elevated anti-dsDNA or extractable nuclear antigen (ENA) antibodies
* Have been on prednisone (or prednisone equivalent) before the screening visit:

  1. at least 8 weeks, and
  2. at a stable dose of 7.5 mg to 30 mg for at least 4 weeks

Exclusion criteria:

A patient is not eligible to participate if he/she:

* Has a history of sensitivity to adrenocorticotropic hormone (ACTH) preparations or porcine products
* Has active lupus nephritis
* Has active central nervous system (CNS) manifestations of SLE

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2016-12-16 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Mallinckrodt
Locations (39):
- United States (16):
  - C.V. Mehta MD Medical Corporation, Hemet, California
  - Inland Rheumatology Clinical Trials, Upland, California
  - Center for Rheumatology Immunology and Arthritis, Fort Lauderdale, Florida
  - San Marcus Research Clinic, Miami, Florida
  - Advanced Pharma CR, Miami, Florida
  - Millennium Research, Ormond Beach, Florida
  - Office of George Timothy Kelly MD, Las Vegas, Nevada
  - NewYork-Presbyterian Columbia University Medical Center, New York, New York
  - DJL Clinical Research, Charlotte, North Carolina
  - Paramount Medical Research & Consulting, Middleburg Heights, Ohio
  - Arthritis & Rheumatology Center of Oklahoma, Oklahoma City, Oklahoma
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - West Tennessee Physicians' Alliance, Jackson, Tennessee
  - Office of Ramesh C. Gupta, MD, Memphis, Tennessee
  - Accurate Clinical Research, Houston, Texas
  - Sun Research Institute, San Antonio, Texas
- Argentina (3):
  - Aprillus Asistencia e Investigación, Buenos Aires
  - Consultorios Médicos Dr. Catalán Pellet, Buenos Aires
  - Centro Medico Privado de Reumatología, San Miguel de Tucumán
- Biomedica Research Group, Santiago, Chile
- Mexico (15):
  - Antiguo Hospital Civil de Guadalajara Fray Antonio Alcalde, Guadalajara, Jalisco
  - IBIOMED Research Unit Aguascalientes, Aguascalientes
  - Centro Especializado en Investigación Clínica, Boca del Río
  - Phylasis Clinicas Research S de RL de CV, Cuautitlán Izcalli
  - Instituto de Investigaciones Aplicadas a la Neurociencia A.C., Durango
  - Unidad de Investigación de las Enfermedades Reumáticas, Mexico City
  - Centro Peninsular de Investigacion Clinica S.C.P., Mérida
  - Köhler and Milstein Research, Mérida
  - Consultorio de Reumatología, México
  - Centro Integral de Reumatologia, México
  - Accelerium Clinical Research, Monterrey
  - Centro de Estudios Clínicos y Especialidades Médicas, Monterrey
  - SMIQ, Querétaro
  - Centro de Alta Especialidad en Reumatologia e Investigación del Potosí, SC, San Luis Potosí City
  - Investigacion Biomedica para el Desarrollo de Farmacos S.A. de C.V., Zapopan
- Peru (4):
  - Investigaciones Clinicas S.A.C. del Instituto de Ginecologia y Reproduccion, Lima
  - Clinica Vesalio, San Borja
  - Hospital de Apoyo Maria Auxiliadora, San Juán de Miraflores
  - Hospital Nacional Cayetano Heredia, San Martín de Porres

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Askanase AD, Wright D, Zhao E, Zhu J, Bilyk R, Furie RA. Post Hoc Biomarker Analyses from a Phase 4, Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial of Repository Corticotropin Injection (Acthar(R) Gel) for Persistently Active Systemic Lupus Erythematosus. Rheumatol Ther. 2021 Dec;8(4):1871-1886. doi: 10.1007/s40744-021-00351-7. Epub 2021 Sep 3. PMID 34478124
- [Derived] Askanase AD, Wan GJ, Panaccio MP, Zhao E, Zhu J, Bilyk R, Furie RA. Patient-Reported Outcomes from a Phase 4, Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial of Repository Corticotropin Injection (Acthar(R) Gel) for Persistently Active Systemic Lupus Erythematosus. Rheumatol Ther. 2021 Mar;8(1):573-584. doi: 10.1007/s40744-021-00294-z. Epub 2021 Mar 9. PMID 33687687
- [Derived] Hannon CW, McCourt C, Lima HC, Chen S, Bennett C. Interventions for cutaneous disease in systemic lupus erythematosus. Cochrane Database Syst Rev. 2021 Mar 9;3(3):CD007478. doi: 10.1002/14651858.CD007478.pub2. PMID 33687069
- [Derived] Askanase AD, Zhao E, Zhu J, Bilyk R, Furie RA. Repository Corticotropin Injection for Persistently Active Systemic Lupus Erythematosus: Results from a Phase 4, Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial. Rheumatol Ther. 2020 Dec;7(4):893-908. doi: 10.1007/s40744-020-00236-1. Epub 2020 Sep 29. PMID 32996096

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 293 who signed informed consent, 172 were randomized into treatment groups
Period: Overall Study
Arm/Group | Placebo Gel | Acthar Gel
Started | 86 | 86
Safety Population | 86 | 86
Modified Intent to Treat (mITT) Populati | 85 | 84
Per Protocol (PP) Population | 72 | 75
Completed Week 16 Visit | 76 | 77
Completed Study Treatment (Week 24) | 73 | 76
Completed (including follow-up) | 71 | 73
Not Completed | 15 | 13
Not completed — Adverse Event | 0 | 4
Not completed — Death | 1 | 0
Not completed — Progressive Disease | 5 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Change of address | 0 | 1
Not completed — Lack of Efficacy | 1 | 0
Not completed — Out of state for indeterminate time | 0 | 1
Not completed — No improvement | 0 | 1
Not completed — Refused follow-up visit | 2 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population (except for study-specific measures)
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Gel | Acthar Gel | Total
Number analyzed (Participants) | 86 | 86 | 172
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.3 (12.99) | 40.1 (12.45) | 39.7 (12.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 76 | 158
  Male | 4 | 10 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 19 | 19 | 38
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 9 | 17
  White | 30 | 33 | 63
  More than one race | 29 | 25 | 54
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Physician's Global Assessment (PGA)
Description: PGA is a 100 mm visual analogue scale where higher scores indicate more severe disease activity. Lower scores indicate improvement.
Time Frame: Baseline, Week 16, Week 24
Population: mITT population with score at the given week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo Gel | Acthar Gel
Number analyzed (Participants) | 85 | 84
score on a scale
  Baseline | 58.8 (15.81) | 60.6 (16.69)
  Week 16: number analyzed (Participants) | 76 | 77
  Week 16 | 33.2 (18.77) | 30.2 (14.89)
  Week 24: number analyzed (Participants) | 73 | 76
  Week 24 | 26.9 (17.76) | 25.5 (17.22)

2. Primary Outcome: British Isles Lupus Assessment Group 2004 (BILAG 2004)
Description: BILAG records disease activity occurring over the past 4 weeks, and is used to determine whether different course of treatment is required. The BILAG-2004 index covers 97 signs/symptoms across 9 organ systems. Each question is answered as 0-not present, 1-improving, 2-same, 3-worse, or 4-new.
  The BILAG-2004 index categorizes disease activity in each organ system into five different levels from A to E. Grade A represents very active disease, Grade B represents moderate disease activity, Grade C indicates mild stable disease, and grade D implies no disease activity, but suggests the organ system had previously been affected. Grade E indicates no current or previous disease activity. A score is applied to each grade of each organ system using coding scheme of A=12, B=8, C=1, and D/E=0 and is summarized as a total score ranging 0-108. Higher scores indicate more severe disease activity.
Time Frame: Baseline, Week 16, Week 24
Population: mITT population with a score at the given week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo Gel | Acthar Gel
Number analyzed (Participants) | 85 | 84
score on a scale
  Baseline | 18.2 (5.15) | 18.0 (5.45)
  Week 16: number analyzed (Participants) | 76 | 77
  Week 16 | 9.7 (6.57) | 7.7 (5.91)
  Week 24: number analyzed (Participants) | 73 | 76
  Week 24 | 8.0 (6.21) | 6.9 (5.87)

3. Primary Outcome: Number of Participants With at Least a 4 Point Change From Baseline in Systemic Lupus Erythematosus Disease Activity Index-2000 (SLEDAI-2K)
Description: The SLEDAI-2K is a modified version of a composite score based on the presence or absence of clinical signs, clinical symptoms, and immunologic laboratory results taken within 10 days of the evaluations. Each of the descriptors has a weighted score and the total score of SLEDAI-2K is the sum of all 24 descriptor scores. The total SLEDAI-2K score falls between 0 and 105, with higher scores representing higher disease activity. Decrease from baseline indicates improvement.
Time Frame: Week 16, Week 24
Population: modified Intent to Treat (mITT)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Gel | Acthar Gel
Number analyzed (Participants) | 85 | 84
Participants
  Week 16 | 40 | 41
  Week 24 | 46 | 44

4. Secondary Outcome: Number of Participants With Severe Flare, Based on the SELENA Flare Index (SFI) at Week 16
Description: Among some adults, having a period of SLE symptoms-called flares-may happen every so often, sometimes even years apart, and go away at other times-called remission. The SFI categorizes SLE flares as mild, moderate or severe.
Time Frame: Week 16
Population: mITT population
Measure: Count of Participants; unit: Participants
Groups:
- Placebo Gel: Participants receive Placebo Gel
- Acthar Gel: Participants receive Acthar Gel
Arm/Group | Placebo Gel | Acthar Gel
Number analyzed (Participants) | 85 | 84
Participants | 3 | 0

5. Secondary Outcome: Mean Cutaneous Lupus Erythematosus Disease Area and Severity Score- Activity (CLASI) Total Activity Score
Description: The CLASI total activity score reflects ongoing inflammation that can be treated, with points given for the presence of erythema, scale, mucous membrane lesions, recent hair loss, and inflammatory alopecia. Mild, moderate, and severe disease correspond with CLASI activity score ranges of 0 to 9, 10 to 20, and 21 to 70, respectively. Higher scores indicate more disease activity, lower scores indicate improvement.
Time Frame: at Baseline and Weeks 4, 8, and 16
Population: mITT population with scores at the given week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo Gel | Acthar Gel
Number analyzed (Participants) | 85 | 84
score on a scale
  Baseline: number analyzed (Participants) | 84 | 82
  Baseline | 7.1 (6.53) | 7.9 (7.48)
  Week 4: number analyzed (Participants) | 82 | 81
  Week 4 | 5.8 (5.57) | 5.6 (5.30)
  Week 8: number analyzed (Participants) | 82 | 78
  Week 8 | 5.0 (5.19) | 5.0 (5.41)
  Week 12: number analyzed (Participants) | 77 | 78
  Week 12 | 4.5 (5.41) | 4.0 (4.08)
  Week 16: number analyzed (Participants) | 75 | 75
  Week 16 | 3.8 (4.36) | 3.4 (3.77)

6. Secondary Outcome: Mean Number of Swollen or Tender Joints on the 28-Joint Count
Description: The 28 Joint Count includes assessment of swelling and tenderness in the shoulders, elbows, wrists, metacarpophalangeal joints, proximal interphalangeal joints and knees. The investigator counts how many of the 28 joints are swollen or tender at the given week.
Time Frame: at Baseline and at Weeks 4, 8, 12 and 16
Population: mITT population with tender and swollen joints at the given week
Measure: Mean (Standard Deviation); unit: Joints
Units Other Than Participants: Joints
Arm/Group | Placebo Gel | Acthar Gel
Number analyzed (Participants) | 85 | 84
Number analyzed (Joints) | 28 | 28
Joints
  Baseline: number analyzed (Participants) | 84 | 81
  Baseline | 7.2 (4.98) | 8.2 (5.85)
  Week 4: number analyzed (Participants) | 82 | 81
  Week 4 | 4.9 (4.77) | 4.2 (4.24)
  Week 8: number analyzed (Participants) | 82 | 78
  Week 8 | 3.8 (4.97) | 2.9 (3.42)
  Week 12: number analyzed (Participants) | 77 | 78
  Week 12 | 2.9 (4.40) | 2.3 (3.00)
  Week 16: number analyzed (Participants) | 75 | 75
  Week 16 | 2.8 (3.67) | 1.9 (3.20)

7. Secondary Outcome: Number of Participants With Decrease in Prednisone Dose to < 7.5 mg/Day at Week 20 and Week 24
Time Frame: Week 20, Week 24
Population: mITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Gel | Acthar Gel
Number analyzed (Participants) | 85 | 84
Participants
  Week 20 | 5 | 3
  Week 24 | 6 | 4

ADVERSE EVENTS:
Time Frame: 24 Weeks
Description: A Treatment-Emergent Adverse Event (TEAE) is defined as an undesirable event that begins or worsens after the first dose of study drug and no later than follow up visit date or no more than 28 days after the last dose of study drug if the follow up visit date is missing. TEAEs were collected in the safety population.
Arm/Group | Placebo Gel | Acthar Gel
All-Cause Mortality (participants affected / at risk) | 1/86 | 0/86
Serious Adverse Events (participants affected / at risk) | 8/86 | 4/86
Other Adverse Events (participants affected / at risk) | 23/86 | 31/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Gel (N=86) | Acthar Gel (N=86)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Soft tissue infection (Infections and infestations) | 1 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 | 2
Drug abuse (Psychiatric disorders) | 1 | 0
Nephrotic syndrome (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Gel (N=86) | Acthar Gel (N=86)
Nasopharyngitis (Infections and infestations) | 6 (6) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 9 (10)
Urinary tract infection (Infections and infestations) | 10 (13) | 6 (6)
Headache (Nervous system disorders) | 5 (6) | 6 (9)
Insomnia (Psychiatric disorders) | 4 (4) | 7 (7)
Hypertension (Vascular disorders) | 0 (0) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-01): https://cdn.clinicaltrials.gov/large-docs/21/NCT02953821/Prot_SAP_000.pdf